CLINICAL TRIAL: NCT00417326
Title: ONO-5046Na Phase II Study - A Pilot Study for Patients With Acute Respiratory Failure
Brief Title: Controlled Study of ONO-5046Na in Patients With Acute Respiratory Failure Associated With Community-Acquired Pneumonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-5046Na-14
Record Dates: First submitted 2006-12-28; First posted 2007-01-01 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Community-acquired Pneumonia
Keywords: ONO-5046Na; acute respiratory failure; community-acquired pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- P (Placebo Comparator)
  Interventions: Drug: ONO-5046Na
- E (Experimental)
  Interventions: Drug: ONO-5046Na

INTERVENTIONS:
Drug: ONO-5046Na — twenty four hour infusion at 0 mg/kg/hr for 14 days
  Arms: P
Drug: ONO-5046Na — twenty four hour intravenous infusion at 0.2 mg/kg/hr for 14 days
  Arms: E

SUMMARY:
The purpose of this study is to determine the safety and efficacy of ONO-5046Na in patients with acute respiratory failure associated with community-acquired pneumonia

ELIGIBILITY:
Inclusion Criteria:

* Patients with community-acquired pneumonia
* Patients with acute respiratory failure

Exclusion Criteria:

* Patients with nosocomial pneumonia
* Patients on mechanical ventilation

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2006-12; Primary Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
pulmonary function | 14 days

SECONDARY OUTCOMES:
mortality | 28 days
ventilator status | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Koji Takehara, Study Director — Ono Pharmaceutical Co. Ltd
Locations (9):
- Japan (9):
  - Chugoku Region, Chugoku
  - Chubu Region, Chūbu
  - Hokkaido Region, Hokkaido
  - Hokuriku Region, Hokuriku
  - Kanto Region, Kanto
  - Kinki Region, Kinki
  - Kyushu Region, Kyushu
  - Shikoku Region, Shikoku
  - Tohoku Region, Tohuku